CLINICAL TRIAL: NCT04473820
Title: Comparison of The Efficacy of Lidocaine-Prilocaine Combination and Vapocoolant Spray to Reduce Pain of IV Cannulation in The Emergency Department: A Randomized Clinical Trial
Brief Title: Comparison of Lidocaine-Prilocaine Combination and Vapocoolant for IV Cannulation Pain in the ED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hadi Mirfazaelian, Assistant Professor of Emergency Medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9111215292
Record Dates: First submitted 2020-07-10; First posted 2020-07-16 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vapocoolant spray (Active Comparator): Patients in this arm will receive vapocoolant spray before IV cannulation.
  Interventions: Drug: Vapocoolant spray
- Lidocaine-Prilocaine cream (Active Comparator): Patients in this arm will receive Lidocaine-Prilocaine cream before IV cannulation.
  Interventions: Drug: Lidocaine-Prilocaine cream

INTERVENTIONS:
Drug: Vapocoolant spray — The spray will be applied continuously from 25 cm distance for less than 5 seconds to the cannulation site.
  Arms: Vapocoolant spray
Drug: Lidocaine-Prilocaine cream — A finger tip (0.5 gr) of the cream will be applied in 4 square cm at cannulation site and will be covered with closed dressing for 45 minutes.
  Arms: Lidocaine-Prilocaine cream

SUMMARY:
Hypothesis: Lidocaine-Prilocaine Combination is as effective as Vapocoolant in treating IV cannulation pain in the emergency department.

DETAILED DESCRIPTION:
Lidocain-Prilocaine combination cream is two amide-type local anesthetics used for topical skin anesthesia. Vapocoolant spray is also another method for providing appropriate analgesia through crayoanesthetic mechanisms. Although there are some contraindications and adverse effects, these are widely used in the Emergency Department (ED) for IV cannulation pain.

ELIGIBILITY:
Inclusion Criteria:

* Low acute patients who are waiting for the admission to the ED and require IV cannulation

Exclusion Criteria:

* Altered mental status
* Uncooperative patients
* Unable to communicate
* Known history of hypersensitivity reaction to cold or amid analgesics
* Analgesic usage in previous 6 hours
* No consent
* Emergent condition
* Pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Cannulation pain: numerical rating score (NRS) | immediately after the procedure.
  The numerical rating score (NRS) will be used for the study. The NRS ranges from 0 (no pain) to 10 (very severe pain). The higher the pain scores the higher the pain severity. The pain severity will be asked from the patients.

SECONDARY OUTCOMES:
Application pain: numerical rating score (NRS) | immediately after the procedure.
  The numerical rating score (NRS) will be used for the study. The NRS ranges from 0 (no pain) to 10 (very severe pain). The higher the pain scores the higher the pain severity. The pain severity will be asked from the patients.
Catheterization attempts | immediately after the procedure.
  Number of times the direction of IV catheter is changed before the successful cannulation. Exit from the skin is also considered an attempt.

CONTACTS AND LOCATIONS:
Locations (1):
- IKCH, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akhgar A, Mazidabadi Farahani A, Akbari H, Sedaghat M, Jalili M, Mirfazaelian H. Comparison of the effects of vapocoolant spray and topical anaesthetic cream (lidocaine-prilocaine) on pain of intravenous cannulation: a randomised controlled trial. Emerg Med J. 2025 May 22;42(6):373-377. doi: 10.1136/emermed-2024-214479. PMID 40118519